CLINICAL TRIAL: NCT06666920
Title: Evaluation of Tooth Color Change and Sensitivity Following Laser-assisted In-office Tooth Bleaching Using Er,Cr:YSGG Laser: a Split-mouth Clinical Study
Brief Title: Er,Cr:YSGG Laser Bleaching on Tooth Color and Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Dimitrios Dionysopoulos, Assistant Professor of the Department of Operative Dentistry of Aristotle University of Thessaloniki, Aristotle University Of Thessaloniki
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 31/23-03-2016
Record Dates: First submitted 2024-10-27; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Tooth Discoloration; Tooth Sensitivity
Keywords: Tooth color change; Laser-assisted tooth bleaching; Spectrophotometer; Tooth sensitivity; Whiteness index
MeSH Terms: conditions — Tooth Discoloration; Dentin Sensitivity | interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Laser-assisted tooth bleaching technique (Experimental): The left hemiarches of the patient's dentition received laser treatment during tooth bleaching procedure
  Interventions: Radiation: laser irradiation
- Conventional tooth bleaching technique (No Intervention): The right hemiarches of the patient's dentition received laser treatment during tooth bleaching procedure

INTERVENTIONS:
Radiation: laser irradiation — Immediately after applying the bleaching agent, the gel on the left upper and lower hemiarches (teeth 21-25 and 31-35) was irradiated using an Er,Cr:YSGG laser (2780 nm). Specifically, an Er,Cr:YSGG solid-state laser device (Waterlase MD Turbo, BIOLASE, Irvine, CA, USA) equipped with a Z-type glass tip (MZ8) measuring 800 μm in diameter and 6 mm in length was used. This tip was attached to the laser system's gold handpiece. The laser parameters for the treatment included an average output power of 1.25 W, a pulse duration of 700 μs (S-mode), and a pulse repetition rate of 10 Hz, without water or air flow, according to a previous study. Each tooth received two 15-s irradiation intervals, one for each 20-min session (totaling 30 s), while maintaining the laser handpiece approximately 2.5 cm from the tooth surface, perpendicular to the enamel. The gel was irradiated using a scanning mode, with the handpiece moved slowly in both horizontal and vertical directions at a speed of 2 mm/s.
  Arms: Laser-assisted tooth bleaching technique

SUMMARY:
The aim of this split-mouth clinical study was to evaluate the tooth color (ΔΕab and ΔΕ00) and whiteness (ΔWID) changes, as well as tooth sensitivity (TS) induced after performing in-office tooth bleaching procedure with or without light-activation of the bleaching gel using Er,Cr:YSGG laser irradiation. Twenty patients with tooth shade A3 or darker were selected for this single-blinded, split-mouth study. The bleaching session was conducted with two 20-min sessions of a 40% hydrogen peroxide bleaching agent assisted by Er,Cr:YSGG laser (2780 nm) irradiation on one side (left) of the maxillary and mandibular teeth and without laser activation on the other hemiarch (right). ΔΕab, ΔΕ00 and ΔWID were evaluated in central incisors and canines using a clinical spectrophotometer immediately, 1 week and 1 month after the bleaching procedure. TS was evaluated pre-operatively and immediately post-operatively using a visual analogue scale (VAS).

DETAILED DESCRIPTION:
The study description adheres to the guidelines of the Consolidated Standards of Reporting Trials (CONSORT) statement. A factorial, single-blind, split-mouth design was employed in this study, with the following factors being examined:

1. Bleaching treatment: two treatment protocols were used, Group 1 (control) - 40% H2O2 bleaching agent and Group 2 - 40% H2O2 bleaching agent + Er,Cr:YSGG laser.
2. Evaluation time: three time points were used for the analysis of bleaching efficacy (T1 at immediately after the treatment, T2 at 7 days after the treatment and T3 at 30 days after the treatment). All color measurements were compared with the baseline values recorded prior to the start of the bleaching treatments. Additionally, tooth sensitivity was assessed at two time points: T1, just before the treatments began, and T2, immediately after the treatments were completed. Patients and the researchers administering the bleaching treatment were not blinded, as it was not possible to conceal whether the bleaching gel was exposed to laser irradiation. However, the evaluator responsible for recording color and sensitivity remained blinded to the treatment conditions.

Bleaching procedure

The study took place at the Postgraduate Dental Clinic of the Department of Operative Dentistry of Aristotle University of Thessaloniki. Initially, twenty volunteers (11 women and 9 men) between the ages of 22 and 48 (mean age 31.1±7.0 years) were enrolled. Patient selection was based on clinical and radiographic examinations, along with a detailed medical history, all conducted prior to the bleaching treatments. Participants were informed about the study's purpose, as well as the potential risks and benefits of the experimental treatment. Those who agreed to participate signed an informed consent form and were provided with both written and verbal instructions regarding hygiene, bleaching gel application, and diet. One week before the tooth bleaching treatment a periodontal treatment using an ultrasonic scaler type Cavitron (KaVo Dental GmbH, Biberach/Riss, Germany) was carried out to remove any external stains or calculus deposits.

All patients received a conventional in-office bleaching treatment using a red-colored bleaching agent with a neutral pH, consisting of 40% H2O2 (Opalescence Boost™ PF 40%, Ultradent Products, Inc., South Jordan, UT, USA). According to the manufacturer's instructions, the contents of the two syringes were blended 25 times and applied in a layer approximately 1 mm thick on the labial surface of the anterior teeth and buccal surface of premolars. After application of a light-cured liquid dam on the gingiva, the bleaching gel was applied on the surface for 20 min, with agitation every 5 min, and subsequently removed using a surgical suction tip. This procedure was repeated for another 20 min (40 min in total) and finally a thorough rinsing with water was followed.

Er,Cr:YSGG laser treatment

Immediately after applying the bleaching agent, the gel on the left upper and lower hemiarches (teeth 21-25 and 31-35) was irradiated using an Er,Cr:YSGG laser (2780 nm). Specifically, an Er,Cr:YSGG solid-state laser device (Waterlase MD Turbo, BIOLASE, Irvine, CA, USA) equipped with a Z-type glass tip (MZ8) measuring 800 μm in diameter and 6 mm in length was used. This tip was attached to the laser system's gold handpiece. The laser parameters for the treatment included an average output power of 1.25 W, a pulse duration of 700 μs (S-mode), and a pulse repetition rate of 10 Hz, without water or air flow, according to a previous study [Dionysopoulos]. Each tooth received two 15-s irradiation intervals, one for each 20-min session (totaling 30 s), while maintaining the laser handpiece approximately 2.5 cm from the tooth surface, perpendicular to the enamel. The gel was irradiated using a scanning mode, with the handpiece moved slowly in both horizontal and vertical directions at a speed of 2 mm/s. This was done to ensure uniform irradiation and complete coverage of the entire surface of the bleaching gel. The fluence for each pulse was 0.45 J/cm², well below the ablation threshold for enamel [Apel]. Each tooth received a total energy of 21.6 J, with an energy delivery rate of 0.72 J/s. To reduce operator variability, the same researcher performed all the whitening procedures.

Evaluation of tooth color and whiteness changes

Color and whiteness changes were evaluated using a spectrophotometer (SpectroShade™, MHT Optic Research AG, Milan, Italy). The measurements were performed at four time points: a) before the bleaching treatment (baseline), b) immediately after the bleaching treatment, c) one week after the bleaching treatment (7 days) and d) one month after the bleaching treatment (30 days). Calibration of the spectrophotometer was carried out at the beginning of each set of measurements using the white and green standards contained in the rechargeable base. Only the center portion of the tooth was used for the collection of data according to Commission Internationale de l'Eclairage Lab (CIELAB) color space. All measurements were repeated twice and averaged under the same light conditions. If ΔΕ between two recordings of the same specimen exceeded 1, new measurements were obtained. The measurements were implemented at room temperature (23±1°C) by the same operator, who did not know which experimental group was measured.

Tooth sensitivity assessment

Tooth sensitivity was analyzed using a visual analog scale (VAS). The scale was represented by a 10 cm horizontal line, limited by two expressions at its ends, with the words "no pain" and "worst pain". Patients were asked about the intensity of spontaneous discomfort caused by the treatment and their responses were scored on the scale, where 0 indicated that patients did not present any painful symptoms and 10 indicated the occurrence of severe sensitivity. When the patient reported sensitivity, they were questioned about the hemiarch in which it occurred, and this information was noted. The values considered on two categories were the percentage of participants who had sensitivity in each treatment group and the intensity of dental sensitivity by treatment group. The analysis between the proportions of patients with sensitivity was performed by Fisher's exact test. The comparison between the intensity of sensitivity on both sides of the split-mouth design was performed by the Mann Whitney test. For both tests, the global level of significance was 95% (α= 0.05).

ELIGIBILITY:
Inclusion Criteria:

* Good overall health
* Healthy oral tissues
* Vital upper and lower anterior teeth
* No carious or non-carious lesions
* Tooth shade A3 or darker

Exclusion Criteria:

* Patients with direct or indirect restorations on their upper or lower anterior teeth.
* Patients using orthodontic appliances.
* Patients undergone previous bleaching treatments.
* Patients with a history of adverse reactions to peroxides.
* Patients taking opioid medications
* Patients having pacemakers.
* Patients with severe tooth discoloration due to tetracycline, trauma, fluorosis, or other causes.
* Patients with clinically verifiable dentin exposure; or those with dental sensitivity or a history of treatment for dental sensitivity.
* Smokers.
* Pregnant or lactating women.
* Patients with neurological disorders.
* Individuals taking medications that could cause photosensitivity.
* Patients with chronic or acute diseases.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Tooth color and whiteness changes | The measurements were performed at four time points: a) before the bleaching treatment (baseline), b) immediately after the bleaching treatment, c) one week after the bleaching treatment (7 days) and d) one month after the bleaching treatment (30 days).
  Tooth color and whiteness changes will be evaluated using a clinical spectrophotometer. According to Commission Internationale de l'Eclairage Lab (CIELAB) color space tooth color change (ΔEab) using the CIELAB system was determined using equation (1):
  ΔEab = [(ΔL)2 + (Δa)2 + (Δb)2]1/2 (1)
  Moreover, tooth color change using the CIEDE2000 system, employing the h (hue) and C (chroma) values was calculated using equation (2):
  ΔE00 = [(ΔL'/KLSL)2 + (ΔC'/KCSC)2 + (ΔH'/KHSH)2 + RT × (ΔC'/KCSC) × (ΔH'/KHSH)]1/2 (2)
  The Whiteness Index for Dentistry (WID) was evaluated based on CIELAB parameters before and after the bleaching treatments, using equations (3) and (4):
  WID= 0.511L - 2.324a - 1.100b (3) ΔWID= WIDi - WID0 (4)

SECONDARY OUTCOMES:
Tooth sensitivity | Measurements were carried out before and immediately after the bleaching procedure
  Tooth sensitivity was analyzed using a visual analog scale (VAS). The scale was represented by a 10 cm horizontal line, limited by two expressions at its ends, with the words "no pain" and "worst pain" (Fig. 1). Patients were asked about the intensity of spontaneous discomfort caused by the treatment and their responses were scored on the scale, where 0 indicated that patients did not present any painful symptoms and 10 indicated the occurrence of severe sensitivity. When the patient reported sensitivity, they were questioned about the hemiarch in which it occurred, and this information was noted. The values considered on two categories were the percentage of participants who had sensitivity in each treatment group and the intensity of dental sensitivity by treatment group.

CONTACTS AND LOCATIONS:
Locations (1):
- Aristotle University of Thessaloniki, Thessaloniki, Central Makedonia, Greece

IPD SHARING:
Plan to Share IPD: Undecided